CLINICAL TRIAL: NCT04910529
Title: The Effect of Yoga Practice on Pain Intensity, Menstruation Symptoms and Quality of Life in Nursing Students With Primary Dysmenorrhea
Brief Title: The Effect of Yoga Practice on Pain Intensity, Menstruation Symptoms and Quality of Life in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Aslıhan Aksu, Research Assistant, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MersinUni
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Primary Dysmenorrhea; Pain, Menstrual; Quality of Life
Keywords: yoga; menstrual pain; menstrual symptoms; quality of life; nursing students; primary dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, two arm, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Participants and the researcher who carried out the application Aslıhan Aksu (A.A.) cannot be blinded due to the nature of the study. When the study is completed, the control and experimental groups will be coded as A and B and the data will be transferred to the computer environment by an independent researcher. The data coded as A and B will be analyzed by a statistician and the findings will be reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga group (Experimental): Hatha yoga, which is one of the most basic yoga methods, will be applied to the students in the study. During each practice within the scope of Hatha yoga, students; breathing exercises, relaxation techniques and warm-up exercises will be applied respectively. In addition to these, asanas (yoga postures) with balance, stretching, relaxation and strengthening components will be applied to the students. This application includes the most basic yoga exercises and does not pose any health risks for practitioners. During the yoga practice in the online environment, the cameras of the students in the yoga group will be turned on and the researcher who has the application will be able to see each student. Yoga will be applied to this group twice a week for 60 minutes each for three menstrual cycles (12 weeks).
  Interventions: Other: Yoga
- Control group (No Intervention): No intervention will be made to the control group, only the data will be collected at the same time as the study group.

INTERVENTIONS:
Other: Yoga — Hatha yoga, which is one of the most basic yoga methods, will be applied to the students in the study. During each practice within the scope of Hatha yoga, students; breathing exercises, relaxation techniques and warm-up exercises will be applied respectively. In addition to these, asanas (yoga postures) with balance, stretching, relaxation and strengthening components will be applied to the students.
  Arms: Yoga group

SUMMARY:
The aim of this randomized controlled study is to evaluate the effect of yoga practice on pain intensity, menstruation symptoms and quality of life in nursing students with primary dysmenorrhea. The hypothesis of this study is that yoga reduces pain and menstrual symptom severity and improves quality of life.

DETAILED DESCRIPTION:
In the study, 52 students will be randomly assigned to intervention (yoga) and control groups. The researcher will provide information about the purpose of the study and the study process by interviewing all the students in the sample online. All students participating in the study, who are in the yoga or control group of the study, will be given a data collection form as a pre-test by the researcher.

Hatha yoga will be applied to the students (n = 26) in the yoga group in the study. Considering the studies conducted with these students, it is planned to practice Hatha yoga for 60 minutes twice a week for three menstrual cycles (12 weeks). Yoga practice will be done online by the researcher Aslıhan Aksu (A.A.), who has a Yoga Alliance-approved yoga instructor certificate, on the determined days and times using appropriate platforms. In the control group (n=26), no intervention will be made for 12 weeks. The results will be collected through data collection forms before the yoga practice and after the 12-week yoga practice is completed. The data collection forms applied to all students in the yoga and control groups at the beginning of the study will be applied to the control group again at the end of 12 weeks. The primary expected result of the study is the effect of yoga on students' menstrual pain intensity. The secondary expected results of the study are to determine the effect of yoga on students' menstrual symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Accepting voluntarily to participate in the study.
* Studying in 1st and 2nd grade between 18 October 2021-16 September 2022 at Mersin University Faculty of Nursing in the Academic Year of 2021-2022,
* Between the ages of 18-24 years,
* Willing to participate in the study,
* Having the facilities (computer, internet, etc.) to participate in the online training,
* Having female gender and a regular menstruation period (occurring at intervals of 21-35 days and lasting 3-8 days),
* Having menstrual pain intensity at least 4 points according to the Visual Pain Scale,
* Having a score of 60 or more according to the Menstruation Symptom Scale,
* Not using hormonal contraception and intrauterine equipment,
* Not pregnant and have not experienced pregnancy before,
* Not having a systemic and chronic disease,
* There is no physical health problem that will prevent/limit yoga practice,
* No diagnosed musculoskeletal disease or no severe heart disease,
* Not practicing yoga regularly,
* No diagnosed psychiatric problems,
* Did not take the Obstetrics-Women's Health and Diseases Nursing course,
* Female students with primary dysmenorrhea who signed the Informed Consent Form.

Exclusion Criteria:

* Not accepting voluntarily to participate in the study.
* Studying in Mersin University Nursing Faculty in the 1st and 2nd grade except 18 October 2021-16 September 2022 in the Academic Year of 2021-2022,
* Younger than 18 years old or over 24 years old,
* Not having the facilities (computer, internet, etc.) to participate in the online training,
* Not having female gender and a regular menstruation period,
* Menstrual pain intensity less than 4 points according to the Visual Pain Scale,
* Having a score of 59 or less according to the Menstruation Symptom Scale,
* Using hormonal contraception and intrauterine device,
* Pregnant and have experienced pregnancy before,
* Having a systemic and chronic disease,
* Having a physical health problem that will prevent/limit yoga practice,
* Diagnosed musculoskeletal disease or severe heart disease,
* Doing regular yoga exercises,
* Having a psychiatric problem,
* Obstetrics-Gynecology and Diseases Nursing course,
* Students without primary dysmenorrhea who do not sign the Informed Consent Form.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Pain will evaluate using The The Short Form of the McGill Pain Questionnaire | Change from before implementation and 12th week of practice
  The main component of the The Short Form of the McGill Pain Questionnaire (SF-MPQ) consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0=none, 1=mild, 2=moderate or 3=severe. In this section, sensory (0-33 points), affective (0-12 points) and total (0-45 points) pain quality scores are obtained. The increase in the total pain scores indicates an increase in the perception of pain. The SF-MPQ also includes the Present Pain Intensity (PPI) Index of the Standard MPQ and a Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Menstrual symptoms will evaluate using the Menstrual Symptom Questionnaire | Change from before implementation and 12th week of practice.
  Menstruation Symptom Scale was developed to evaluate menstrual pain and symptoms. Participants in the scale give a value between 1 and 5 (1 = never, 2 = sometimes, 3 = occasionally, 4 = often, 5 = always) to symptoms they experience about menstruation. Scores ranging from 20 to 80 points are obtained in the scale. Increasing the average score indicates that the severity of menstrual symptoms increased.
Quality of life will evaluate using SF-36 Quality of Life Questionnaire | Change from before implementation and 12th week of practice
  SF-36 Quality of Life Questionnaire covers many concepts related to general health and is used frequently today. SF-36 consists of 8 sub-dimensions (physical function, physical role restriction, emotional role restriction, bodily pain, general health perception, energy / vitality, social function, mental health) and 36 questions in total. In the scale, eight sub-dimensions can be evaluated separately as well as in two main dimensions, physical and mental dimensions. Subscales evaluate health between 0 and 100 points (0 point = bad health, 100 points = good health).

CONTACTS AND LOCATIONS:
Overall Officials: Duygu VEFİKULUCAY YILMAZ, PhD, Study Director — Professor
Locations (1):
- Mersin University, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No